CLINICAL TRIAL: NCT01796847
Title: Influence of PTEN on Glycemic Variability and Clinical Outcome in the Critically Ill Patient.
Brief Title: Relationship Between PTEN and Glycemic Variability and Outcome in Critically Ill Patients
Acronym: GLUPTEN
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Laviano, Associate Professor, University of Roma La Sapienza
Other Study IDs: LAVPTEN
Record Dates: First submitted 2013-02-11; First posted 2013-02-22 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Critical Illness; Hyperglycemia
Keywords: ICU; Hyperglycemia; Length of stay
MeSH Terms: conditions — Critical Illness; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PTEN, hyperglycemia

SUMMARY:
Glycemic variability in critically ill patients is a recognized negative prognostic factor. The molecular mechanisms determining inter-patients variability in glucose metabolism during stress are not fully understood. The Phosphatase and Tensin homolog (PTEN) is known to influence glucose homeostasis by interfering in intracellular insulin signaling.

Aim of this study is to ascertain whether differential expression of PTEN in critically ill patients correlates with glycemic variability and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* trauma
* provision informed consent

Exclusion Criteria:

* diabetes
* impaired fasting glucose levels

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Truma patients admitted to general ICU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Length of ICU stay | Day 1 up to day 28

SECONDARY OUTCOMES:
Glycemic variability as expressed by standard deviation of the glycemia measurements | Day 1 up to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Laviano, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- University of Rome La Sapienza, University Hospital, Rome, Italy

REFERENCES:
- [Derived] Molfino A, Alessandri F, Mosillo P, Dell'Utri D, Farcomeni A, Amabile MI, Laviano A. PTEN expression and its association with glucose control and calorie supplementation in critically ill patients. Clin Nutr. 2018 Dec;37(6 Pt A):2186-2190. doi: 10.1016/j.clnu.2017.10.021. Epub 2017 Nov 4. PMID 29154111